CLINICAL TRIAL: NCT03174587
Title: A Phase 1 Study to Evaluate the Safety of CS20AT04 Inj. in Subjects With Lupus Nephritis.
Brief Title: Evaluate the Safety of CS20AT04 Inj. in Subjects With Lupus Nephritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corestemchemon, Inc. (Industry)
Collaborators: Hanyang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS20AT04-LN101
Record Dates: First submitted 2017-05-31; First posted 2017-06-02 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Lupus Nephritis
Keywords: Systemic lupus erythematosus; HLA-haplo-matching; allogenic bone marrow derived mesenchymal stem cell; Phase 1 clinical trial
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CS20AT04 (Experimental): Test group : CS20AT04 (allogenic bone marrow derived mesenchymal stem cells.)
  Interventions: Biological: allogenic bone marrow derived mesenchymal stem cells

INTERVENTIONS:
Biological: allogenic bone marrow derived mesenchymal stem cells — Step -1 dose : 1.0x10^6cells/kg Step 1 dose : 2.0x10^6cells/kg Step 2 dose : 3.0x10^6cells/kg The single injection of CS20AT04 Inj. in the peripheral veins.(IV) The duration of follow up study following the single dose of CS20AT04 is 28 days
  Other Names: CS20AT04

SUMMARY:
The purpose of conducting phase 1 trial to evaluate the safety and tolerability of allogenic bone marrow-derived mesenchymal stem cells(CS20AT04) in subjects with lupus nephritis.

Evaluating DLT by IV injection according to dose-escalating in lupus nephritis patients.

DETAILED DESCRIPTION:
Lupus is a representative autoimmune disease that affects the whole body. It is occurred by generation of autoantibody and immune complex due to abnormal activation of the immune cells on the basis of abnormal immune responses.

Although about 50% of lupus patients have lupus nephritis, there is no therapy product targeted for the lupus nephritis now.

We have performed the pre-clinical and clinical studies using allogenic bone marrow derived mesenchymal stem cells in SLE.

CS20AT04 has anti-inflammatory effects, controls activity of immune cells and reduces generation of autoantibodies. So, it is expected to have treatment effects of lupus nephritis.

The clinical trial was designed as a single center, open-label, phase 1 clinical trials.

If that subject's written informed consent form to participate in this clinical trial will be conducted the required examinations and tests in accordance with the study protocol within 56 days investigational drug administration.

Then, the register for each dose step. For the final 3 subjects in the inclusion / exclusion criteria and be administered a drug test.

Check the adverse events for more than four hours after administration of the investigational drug, and will determine whether the expression of adverse drug reaction(ADR) by the visit after 3 days, 7 days and 28 days.

Except for dose administration, all subject are tested in the same schedule. As a result of evaluating severity of AE divided into grades in accordance with the CTCAE (Version 4.0) standards.

ELIGIBILITY:
Inclusion Criteria:

* Male and female Patients aged ≥18 years and < 70years.
* Patients with HLA-haplo-matched bone marrow donor is less than 70 years old.
* Clinical diagnosis of SLE by American College of Rheumatology (ACR) criteria.
* Patients had suffered from active renal disease in the past or patients has active renal disease now. Active renal disese should have include below.

  1. Spot urine protein/creatinine ratio ≥ 1.0 and ① >5 RBC/HPF, ② >5 WBC/HPF, ③ columnar cell.
  2. Biopsy confirmed active type III or type IV, or type V lupus nephritis.
* Patients can be immunosuppressive agent to , steroids, taking, such as anti-Malarials (hydroxychloroquine) in a certain capacity, during the test period, to maintain the same capacity before 4-weeks screening.
* Patients who consented to participate in the study in writing by themselves or their legal representatives.

Exclusion Criteria:

* Those who do not kidney disease for SLE.
* Patients with a history of hypersensitivity, such as heavy metal poisoning similar to drug testing and drug ingredients.
* Patients a history Major organs (kidney, liver, lung, heart) transplant or liver hematopoietic cells / transplant or during of scheduled transplantation clinical trial.
* patients a history of kidney dialysis or during of the scheduled dialysis clinical trials within 2 weeks prior to the screening.
* Tested positive for hepatitis B(HBsAg, Anti-HBcAB, HBV-DNA) and hepatitis C(Anti-HCV, HCV-RNA) \.
* Patients a history of anaphylactic reaction for the parenteral administration of a monoclonal antibody or contrast agent, a mouse protein or human.
* Patients whose e-GFR ≤ 30mL/min at screening.
* Patients with a history of malignancy within 5 years prior to the screening(basal cell carcinoma of skin, squamous cell carcinoma of skin, or cervical intraepithelial neoplasia are excluded).
* Patients who were administered drug of the follow within 6 months prior to the screening.

  * nitrogen mustard, chlorambucil, vin·cris·tine, procarbazine, Abatacept, Rituximab, Belimumab
* Patients who were administered drug of the follow within 3 months prior to the screening.

  * Anti-TNF therapy(Etanercept, adalimumab, Infliximab, golimumab, Tocilizumab)
  * Interleukin-1 receptor antagonist(anakinra)
  * Intravenous immunoglobulin(IVIG)
  * Plasmapheresis
* Those who are hypersensitive to antibiotics including penicillin and streptomycin.
* Patients with systemic infection at screening.
* Uncontrolled hypertension or diabetes.
* If that may affect proteinuria increased capacity or begin taking medication(ACE inhibitors, ARB (Angiotensin Receptor Blocker)) (However, more than four weeks allowed capacity, taking is possible during the trial period without changing capacity).
* Patients who showed myocardial infarction or angina on ECG at screening, or received stent procedure or bypass.
* Patients who were administered another study drug 3 months prior to the study.
* Patients with severe mental disease(for example, schizophrenia, bipolar disorder etc;).
* Patients are expected to be administered the combination contraindicated drugs about inevitable or taker within clinical trial.
* Women of childbearing age are not implement adequate contraception during clinical trials. the proper method of contraception, which has Oral contraceptive continued more than four weeks, a surgical procedures including the insertion loop, condom use etc. and Medically it is determined that there is no possibility of pregnant women do not belong to women of childbearing age due to the ovary removal, hysterectomy and menopause, etc.
* Pregnant women or nursing women.
* Except as permitted in the following Case and laboratory test results than moderate adverse events(NCI-CTC (National Cancer Institute-Common Toxicity Criteria) version 4.0) grade 3.

  * proteinuria
  * hematuria
  * pyuria
  * Columnar
  * Hypoalbuminemia caused by lupus nephritis
  * Class III due to stable prothrombin time of warfarin therapy
  * Lupus anticoagulant group, and are not associated with liver disease or stable anticoagulation 3 grade partial thromboplastin time
  * Lupus due to hepatitis and alcoholic liver disease, are not associated with uncontrolled diabetes or viral hepatitis stable 3 grade gamma glutamyl transferase (GGT) increases. If it appears to be less than ALT and / or AST is above all on the second level.
  * Stable grade 3 neutropenia or white blood cell count
* Patients who previously received stem cell therapy.
* Subjects who by the investigator to make them ineligible for participation in this clinical study.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2019-08-19 (Actual)

PRIMARY OUTCOMES:
Safety assessment(evaluation) | 28 days after administration
  Adverse events(AE), Laboratory test(hematology/blood chemistry, urine test), Vital signs, Physical examination, ECG

CONTACTS AND LOCATIONS:
Overall Officials: SANG-CHEOL BAE, Principal Investigator — Hanyang University
Locations (1):
- Hanyang university hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jang E, Jeong M, Kim S, Jang K, Kang BK, Lee DY, Bae SC, Kim KS, Youn J. Infusion of Human Bone Marrow-Derived Mesenchymal Stem Cells Alleviates Autoimmune Nephritis in a Lupus Model by Suppressing Follicular Helper T-Cell Development. Cell Transplant. 2016;25(1):1-15. doi: 10.3727/096368915X688173. Epub 2015 May 13. PMID 25975931
- [Background] Shim JS, Sung YK, Joo YB, Lee HS, Bae SC. Prevalence and incidence of systemic lupus erythematosus in South Korea. Rheumatol Int. 2014 Jul;34(7):909-17. doi: 10.1007/s00296-013-2915-9. Epub 2013 Dec 10. PMID 24322455
- See also: Corestem Inc. — http://www.corestem.com